CLINICAL TRIAL: NCT05679128
Title: Palpation Versus Ultrasonography for Identifying the Cricothyroid Membrane in Case of a Laterally Deviated Larynx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, Head of Airway Management development, Consultant anaesthesiologist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Devtrach1
Record Dates: First submitted 2022-11-17; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Airway Management

STUDY DESIGN:
Intervention Model Description: randomised to either "palpation" or "ultrasonography"
  The participants are thus arandomised to use either "palpation" or to use "ultrasonography" to DIAGNOSE the position of the cricothyroid membrane
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palpation (Active Comparator): digital palpation used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: identification of the cricothyroid membrane using Palpation
- ultrasonography (Experimental): Ultrasonography used to identify the cricothyroid membrane
  Interventions: Diagnostic Test: Identification of the cricothyroid membrane using ultrasonography

INTERVENTIONS:
Diagnostic Test: identification of the cricothyroid membrane using Palpation — identification of the cricothyroid using PALPATION, a procedure used to prepare for front of neck airway access
  Arms: palpation
Diagnostic Test: Identification of the cricothyroid membrane using ultrasonography — identification of the cricothyroid membrane, using ULTRASONOGRAPHY, a procedure used to prepare for front of neck airway access
  Arms: ultrasonography

SUMMARY:
test persons, anaesthesiologists will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography. The larynx-model is deviated to one of the sides to simulate a patient with neck pathology

DETAILED DESCRIPTION:
test persons, anaesthesiologists will identify the cricothyroid membrane on a silicone model of the neck with either palpation or ultrasonography. The larynx-model is deviated to one of the sides to simulate a patient with neck pathology.

The test persons are randomised to use other palpation or ultrasonography. Al attempts are video-taped

ELIGIBILITY:
Inclusion Criteria:

* Participants in a course of airway management

Exclusion Criteria: unwillingness to participate

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Correct identification of the cricothyroid membrane within a minute | 1 minute
  The fraction of identifications of the location of the cricothyroid membrane made by the participants, that is actually correct. ie the succesrate of correct identification.

SECONDARY OUTCOMES:
Time taken to identification of the estimated location of the cricothyroid membrane. | up to 3 minutes
  The time elapsing from the participants initiate their attempt at identificating the cricothyroid membrane until they have finished their attempt at identifying the cricothyroid membrane.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lohse R, Wagner N, Kristensen MS. Palpation Versus Ultrasonography for Identifying the Cricothyroid Membrane in Case of a Laterally Deviated Larynx: A Randomized Trial. Anesth Analg. 2024 Jul 1;139(1):195-200. doi: 10.1213/ANE.0000000000006867. Epub 2024 Jan 31. PMID 38295131